CLINICAL TRIAL: NCT03165357
Title: The Effect of Sodium Bicarbonate Supplementation on Physical Capacity and Body Composition in Trained Athletes
Brief Title: Sodium Bicarbonate Supplementation in Athletes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of PhysED (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ULS00002
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Supplementation; Sport
Keywords: Crossfit; Sodium bicarbonate; Physical capacity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium bicarbonate (Experimental): Group taking oral NaHCO3 supplementation in a progressive-dose regimen.
  Interventions:
  The experimental procedure for each athlete included a 10-day NaHCO3 supplementation in a progressive-dose regimen in order to reduce the likelihood of gastrointestinal side effects (from 37.5 to 150 mg ∙ kg-1). NaHCO3 was administered in the form of unmarked disk-shaped tablets (Alkala T, SANUM, Poland). The tablets were ingested with at least 250 mL of water and could be either swallowed or dissolved in the mouth. On training days the supplements were taken in the morning, in the evening and 1.5 hours before training session. On rest days the supplements were taken in the morning, in the afternoon and in the evening.
  Between the 10-day NaHCO3 and PLA or a PLA and NaHCO3 treatments, a 14-day washout period was introduced.
  Interventions: Dietary Supplement: Sodium bicarbonate supplementation
- Placebo (maltodextrin) (Placebo Comparator): Group taking oral supplementation with placebo (maltodextrin).
  Interventions:
  The experimental procedure for each athlete included a 10-day placebo administration. Placebo was ingested with at least 250 mL of water. On training days the supplements were taken in the morning, in the evening and 1.5 hours before training session. On rest days the supplements were taken in the morning, in the afternoon and in the evening.
  Between the 10-day NaHCO3 and PLA or a PLA and NaHCO3 treatments, a 14-day washout period was introduced.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate supplementation
  Arms: Sodium bicarbonate
Dietary Supplement: Placebo treatment
  Arms: Placebo (maltodextrin)

SUMMARY:
The purpose of this study was to verify the effect of 10-day sodium bicarbonate (NaHCO3) and placebo (PLA) supplementation on body composition, physical capacity, as well as concentrations of the selected biochemical blood markers in trained athletes, in a randomised, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Sodium bicarbonate (NaHCO3) was proposed as an ergogenic agent, because it improves high-intensity and resistance exercise performance. Until now the major limitation to NaHCO3 supplementation has been the gastrointestinal (GI) side effects. Therefore, this study aims to examine the effect of chronic, progressive- dose NaHCO3 ingestion on physical capacity, body composition and concentrations of the selected biochemical blood markers in trained athletes, in a randomised, double-blind, placebo-controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* a current medical clearance to practice sports,
* training experience: at least 2 years (of CrossFit training),
* minimum of 3 workout sessions (CrossFit) a week,
* 20-43 years.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol.

Ages: 20 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Changes in aerobic capacity after sodium bicarbonate supplementation | Baseline and after 10 days
  The incremental cycling test (ICT)
Changes in specific performance capacity after sodium bicarbonate supplementation | Baseline and after 10 days
  The CrossFit-specific physical fitness test: Fight Gone Bad (FGB)

SECONDARY OUTCOMES:
Changes in fat mass and fat free mass after sodium bicarbonate supplementation | Baseline and after 10 days
  Fat mass (kg) and fat free mass (kg) analysis
Changes of red and white blood cell concentration in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Red blood cells (RBC) [mln/mm³] and white blood cells (WBC) [mln/mm³] concentration analysis
Changes in blood glucose and hemoglobin concentration after sodium bicarbonate supplementation | Baseline and after 10 days
  Hemoglobin (Hb) [g/dl] and glucose [g/dl] concentration analysis
Changes in blood hematocrit levels after sodium bicarbonate supplementation | Baseline and after 10 days
  Hematocrit (HCT) [%] level analysis
Changes of lactate and pyruvate concentration in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Lactate [mmol/L] and pyruvate [mmol/L] concentration analysis
Changes of creatine kinase and lactate dehydrogenase activity in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Creatine kinase [U/L] and lactate dehydrogenase [U/L] activity analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jeszka, Professor, Study Chair — Department of Hygiene and Human Nutrition, Poznan University of Life Sciences, Poznan, Poland
Locations (1):
- Poznan University of Life Sciences, ul.Wojska Polskiego 31, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level recorded indicators (body composition, aerobic and anaerobic capacity indicators, levels of biochemical markers), without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal